CLINICAL TRIAL: NCT02904161
Title: Detection of Circulating Tumor Cells in Peripheral Blood From Healthy Volunteers and Patients With Cancer
Status: Completed | Type: Observational
Sponsor: MiCareo Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MCPZ12001J1
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-09

CONDITIONS: Circulating Tumor Cells (CTCs)
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- first stage: For the first stage, 60 healthy volunteers, 10 patients with stage 4 breast cancer and 10 patients with other types of cancer will be recruited.
- second stage: For the second stage, approximately 65 breast cancer patients will be recruited.

SUMMARY:
To address the challenges of isolating and analyzing rare cells, this study aims to validate technical diagnostic instrumentation, tests, protocols and analysis to correlate the number of circulating tumor cells present in whole blood for predicting cancer prognosis and treatment efficacy. Investigators propose to enroll and follow cohorts of cancer patients. Blood samples will be collected from these patients at regular intervals as determined by their doctors. The patient's disease progression will be monitored over the lifetime of this study. The specific aims are to isolate, enumerate and analyze the number of circulating tumor cells (CTCs) in patient blood using chip-based sorting, filtration and imaging techniques. Investigators will also use this study to optimize diagnostic instrumentation, test protocols and downstream CTC analysis. Investigators may also correlate the results of these tests with the prognosis of the patients as well as any clinical evidence (e.g. from radiological imaging scans). While investigators focus on prognosis in this study, these correlated tests potentially may also be valuable in future studies for early diagnosis and monitoring of cancer.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the first stage of the study, subjects must fulfill all of the following criteria:

1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Patients diagnosed with stage 4 breast cancer or other types of cancer or chosen to be part of one of the negative control population cohorts.

For inclusion in the second stage of the study, subjects must fulfill all of the following criteria:

1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Patients diagnosed with breast cancer or other types of cancer or chosen to be part of one of the negative control population cohorts.

Exclusion Criteria:

The following is regarded as a criterion for exclusion from the study and applicable to both 2 stages :

1. Subject has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers and breast cancer patients
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2012-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided